CLINICAL TRIAL: NCT05906121
Title: Lidocaine and Ketamine Levels in Plasma After Simultaneous Lidocaine/Ketamine Infusions. An Observational Assessment of Therapy Effects and Side-effects.
Brief Title: Lidocaine and Ketamine Levels in Plasma After Simultaneous Lidocaine/Ketamine Infusions
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-00658; am23Schneider2
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Chronic Pain
Keywords: Lidocaine; Ketamine; lidocaine/ketamine infusions; Short form - McGill Pain Questionnaire (SF - MPQ); Beck Depression Questionnaire (BDI-II)
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: lidocaine-ketamine infusions — Lidocaine and ketamine are infused over a period of 30 minutes. The dosage of lidocaine is 4mg/kg is maintained throughout the infusions, and the dosage of ketamine is increased within the first three infusions from 0.15mg/kg at the first, to 0.25mg/kg at the second and 0.5mg/kg at the third infusion. In case patients already experiencing sufficient analgesic effect and/or improvement in quality of life after the 1st or 2nd infusion or if side effects do not allow a further dose increase, no further step up of ketamine dosage is made. As a part of this study, at the end of the first, second and third infusion, side effects will be screened using customized questionnaires (SF - MPQ, BDI-II)

SUMMARY:
The aim of this monocentric observational pilot study is to measure the lidocaine plasma level in a limited number of patients to generate explorative data on inter- and intrapersonal stability and safety of drug plasma levels and to investigate whether higher plasma levels of ketamine can be correlated with a better analgesic effect.

DETAILED DESCRIPTION:
There are different treatment strategies for chronic pain. One possible treatment strategy, especially for therapy-resistant pain, is intravenous infusions with certain pharmacological agents, such as lidocaine and ketamine. This study is to measure the concentration of lidocaine in the plasma of patients at the University Hospital of Basel (USB) after an intravenous infusion with 4mg/kg lidocaine over 30 minutes in order to generate explorative data on inter- and intrapersonal stability and safety of drug plasma levels. The prospective side effects of lidocaine and ketamine is assessed and the plasma levels are correlated with the analgesic efficacy and change in possible depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Patient is a new recipient of lidocaine-ketamine infusions
* Patient is able to provide Informed Consent

Exclusion Criteria:

* Contraindication to blood sampling (on arm not used for infusion)
* Insufficient knowledge of German language
* Inability to give consent
* Patient is under 18 years of age
* Contraindication to treatment with lidocaine and/or ketamine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 15 patients (10 + Drop-out of 50%) newly receiving lidocaine-ketamine infusions at the USB will be randomly selected.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2023-05-16 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Change in Lidocaine plasma level | After infusion 1 (Baseline), after infusion 2 (28 days after infusion 1), after infusion 3 (28 days after infusion 2)
  Concentration of lidocaine in the plasma of patients who received an intravenous infusion with 4mg/kg lidocaine and 0.15 - 0.5mg/kg ketamine over 30 minutes at the time directly after the infusion.

SECONDARY OUTCOMES:
Change in Ketamine plasma level | After infusion 1 (Baseline), after infusion 2 (28 days after infusion 1), after infusion 3 (28 days after infusion 2)
  Concentration of ketamine in the plasma of patients who received an intravenous infusion with 4mg/kg lidocaine and 0.15 - 0.5mg/kg ketamine over 30 minutes at the time directly after the infusion.
Change in pain assessment | After infusion 1 (Baseline), after infusion 2 (28 days after infusion 1), after infusion 3 (28 days after infusion 2)
  Change of pain assessed by the Short form - McGill Pain Questionnaire (SF- MPQ). he main component of the SF-MPQ consists of 15 descriptors (11 sensory; 4 affective) which are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate or 3 = severe.
Change in mood assessment | After infusion 1 (Baseline), after infusion 2 (28 days after infusion 1), after infusion 3 (28 days after infusion 2)
  Change of mood assessed by the Beck Depression Questionnaire II (BDI-II); Conventional cutoffs are 0-9 for normal range, 10-18 for mild to moderate depression, 19-29 for moderate to severe depression, and 30-63 for severe depression

CONTACTS AND LOCATIONS:
Overall Officials: Wilhelm Ruppen, Prof., Principal Investigator — Department of Anaesthesiology, University Hospital of Basel (USB)
Locations (1):
- Department of Anaesthesiology, University Hospital of Basel (USB), Basel, Switzerland

DOCUMENTS (1):
  • Study Protocol (2023-05-02): https://cdn.clinicaltrials.gov/large-docs/21/NCT05906121/Prot_000.pdf